CLINICAL TRIAL: NCT01487460
Title: A First-in-human Randomized, Double-blind, Placebo-controlled, 4-part Study to Assess Safety, Tolerability, Pharmacokinetics (Including Open Label Study of Food Effect and Interaction With Simvastatin) and Pharmacodynamics of Interwoven Single- and Multiple-ascending Doses of TAP311 in Healthy Subjects and Dyslipidemic Patients.
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of TAP311 in Healthy Subjects and Dyslipidemic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CTAP311X2101
Record Dates: First submitted 2011-11-28; First posted 2011-12-07 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2016-04

CONDITIONS: Dyslipidemia; Healthy Volunteers
Keywords: High cholesterol levels; Hyperlipidemia; High-density Lipoprotein; Low-density Lipoprotein; Simvastatin
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- TAP311 in Healthy Volunteers (Experimental)
  Interventions: Drug: TAP311
- Matching Placebo (Placebo Comparator): Healthy Volunteers and Patients will be treated in Placebo group.
  Interventions: Drug: TAP311
- TAP311 and Simvastatin (Experimental)
  Interventions: Drug: TAP311
- TAP311 in Patients (Experimental)
  Interventions: Drug: TAP311

INTERVENTIONS:
Drug: TAP311

SUMMARY:
This study will assess the safety, tolerability, and effect of TAP311 on blood lipids in healthy subjects and in patients who have dyslipidemia. The effect of food on TAP311 concentration in blood and effect of TAP311 administration on simvastatin concentration will also be assessed in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects age 18 to 65 years of age included, and in good health as determined by past medical history, physical examination, electrocardiogram, and laboratory tests at screening.
* OR untreated dyslipidemic patients.
* Subjects must weigh at least 50 kg to participate in the study, and must have a body mass index (BMI) within the range of 18 - 36 kg/m2.
* Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion Criteria:

* Use of other investigational drugs at the time of enrollment.
* Active treatment for type 1 diabetes or type 2 diabetes mellitus.
* A past medical history of ECG abnormalities, documented cardiac arrhythmias or cardiovascular diseases.
* History of malignancy of any organ system, treated or untreated, within the past 5 years.
* Pregnant or nursing (lactating) women.
* Smokers.
* Use of any prescription drugs, herbal supplements and/or over-the-counter (OTC) medication, dietary supplements.
* History of drug or alcohol abuse within the 12 months prior to dosing.
* Any surgical or medical condition, acute or unstable chronic disease which may, based on the investigator's opinion, jeopardize the patient in case of participation in the study

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2011-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple doses of TAP311 in healthy subjects and patients with dyslipidemia | Up to 21 days
  Number of patients with adverse events and changes from baseline in vital signs, ECG and clinical labs (blood chemistry, hematology and urinalysis).

SECONDARY OUTCOMES:
TAP311 concentrations in blood and urine following administration of single and multiple doses in healthy subjects and in patients with dyslipidemia. | 25 timepoints over 17 days
Effect of TAP311 administration on simvastatin (and metabolite) blood concentration in healthy subjects. | 10 days
  Simvastatin (and metabolite) blood concentration before and after TAP311 treatment.
Effect of food on TAP311 blood concentration in healthy subjects. | 3 days
  TAP311 blood concentration when the drug is administered with and without food.
Effects of TAP311 on total cholesterol in patients with dyslipidemia | 8 timepoints over 15 days
  Total cholesterol blood concentration before and after TAP311 treatment.
Effects of TAP311 on Low Density Lipoprotein (LDL-C) in patients with dyslipidemia | 8 timepoints over 15 days
  LDL-C blood concentration before and after TAP311 treatment.
Effects of TAP311 on high density lipoprotein (HDL-C)in patients with dyslipidemia. | 8 timepoints over 15 days
  HDL-C blood concentration before and after TAP311 treatment.
Effects of TAP311 on triglycerides in patients with Dyslipidemia | 8 timepoints over 15 days
  Triglycerides concentration in blood before and after TAP311 treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Miramar, Florida, United States

REFERENCES:
- See also: Results for CTAP311X2101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=9083